CLINICAL TRIAL: NCT03162367
Title: Comparison Study OF Efficacy Of Autologous Epidermal Cell Suspension And Silver Sulfadiazine Ointment In Second Degree Burn
Brief Title: Efficacy Of Autologous Epidermal Cell Suspension And Silver Sulfadiazine Ointment In Burn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCARM Institute, Tabriz, Iran (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCARM-Skin-002
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2019-06

CONDITIONS: Burn
Keywords: Burn; Epidermal cell suspension
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous epidermal cell suspension group (Experimental)
  Interventions: Biological: Autologous epidermal cell suspension
- Silver sulfadiazine ointment group (Active Comparator)
  Interventions: Drug: Silver sulfadiazine ointment

INTERVENTIONS:
Biological: Autologous epidermal cell suspension — First skin samples taken from normal skin by 4mm punch will be send to laboratory for preparation of epidermal cell suspension and this suspension transfer to one area of second degree burn
  Arms: Autologous epidermal cell suspension group
Drug: Silver sulfadiazine ointment — the area with second degree burn dresses by silver sulfadiazine ointment and dressing change each 12 hour till 10 day
  Arms: Silver sulfadiazine ointment group

SUMMARY:
Different medical treatments are available for treatment of skin burns such as skin grafts and silver sulfadiazine ointment. These treatments are used for second degree burn as routine technique in burns units. Cell therapy is a new approach for treatment of skin disease.In this study we use autologous epidermal cell suspension to achieve better cosmetic and functional results in treatment of second degree burn.

DETAILED DESCRIPTION:
In this study 20 patients in Burn Department of Sina Hospital Tabriz, with at least 2 areas of second degree burn randomly choose. First skin samples are taken from normal skin by 4mm punch and send to the laboratory for preparation of epidermal cell suspension and this suspension is transferred to the one area of second degree burn in each patient and the other area in the same patient dresses by silver sulfadiazine ointment. The dressing changes are followed up for 12h for first assessment of therapy until 10th day after intervention. In the days of 5, 10, 15 and 20 the percentage of re-epithelization for each treatment will be measured. After 2 months, patients are visited and any complications check for scar formation, pain, post inflammatory hyper-pigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient with second degree burn admitted in burn unit

Exclusion Criteria:

* Pregnancy-lactation
* Immunosuppression like receiving chemotherapy or radiotherapy
* Patient unsatisfied to going on study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in re-epithelization rate with autologous epidermal cell suspension graft from Baseline | up to 20 days
  Measurement the percentage of re-epithelization ( 0-30%=poor; 30-60%=moderate; 60-90%=good; >90%=complete)
Change in re-epithelization rate with silver sulfadiazine ointment from Baseline | up to 20 days
  Measure percentage of re-epithelization ( 0-30%=poor; 30-60%=moderate; 60-90%=good; >90%=complete)

SECONDARY OUTCOMES:
Scar formation | After 2 month
  Observe patient and take photo
Post inflammatory hyperpigmentation | After 2 month
  Observe patient and take photo

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Reza Ranjkesh, MD, Dermatologist, Study Director — SCARM institute
Locations (1):
- Sina hospital, Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] You HJ, Han SK. Cell therapy for wound healing. J Korean Med Sci. 2014 Mar;29(3):311-9. doi: 10.3346/jkms.2014.29.3.311. Epub 2014 Feb 27. PMID 24616577
- [Result] Zhao H, Chen Y, Zhang C, Fu X. Autologous epidermal cell suspension: A promising treatment for chronic wounds. J Tissue Viability. 2016 Feb;25(1):50-6. doi: 10.1016/j.jtv.2015.11.003. Epub 2015 Dec 8. PMID 26706649
- [Result] Mcheik JN, Barrault C, Levard G, Morel F, Bernard FX, Lecron JC. Epidermal healing in burns: autologous keratinocyte transplantation as a standard procedure: update and perspective. Plast Reconstr Surg Glob Open. 2014 Oct 7;2(9):e218. doi: 10.1097/GOX.0000000000000176. eCollection 2014 Sep. PMID 25426401
- [Result] Gardien KL, Marck RE, Bloemen MC, Waaijman T, Gibbs S, Ulrich MM, Middelkoop E; Dutch Outback Study Group1. Outcome of Burns Treated With Autologous Cultured Proliferating Epidermal Cells: A Prospective Randomized Multicenter Intrapatient Comparative Trial. Cell Transplant. 2016;25(3):437-48. doi: 10.3727/096368915X689569. Epub 2015 Sep 28. PMID 26419871